CLINICAL TRIAL: NCT02750501
Title: Absorption and Safety With Sustained Use of RELiZORB Evaluation (ASSURE) Study in Patients With Cystic Fibrosis Receiving Enteral Feeding
Brief Title: Absorption and Safety With Sustained Use of RELiZORB Evaluation (ASSURE) Study
Acronym: ASSURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcresta Therapeutics, Inc. (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 0000498-02
Record Dates: First submitted 2016-04-20; First posted 2016-04-25 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-06

CONDITIONS: Cystic Fibrosis
Keywords: CF, EPI, diabetes, PERT, LCPUFA, DHA, EPA, Omega-3 index
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm: Open label RELiZORB Cartridge & Impact Peptide 1.5 (Other): RELiZORB (immobilized lipase) cartridge and Impact Peptide 1.5 with enteral feedings ranging from 500 mL to 1,000 mL per feeding for a period of 90 days.
  Interventions: Device: RELiZORB (immobilized lipase) cartridge; Other: Impact Peptide 1.5

INTERVENTIONS:
Device: RELiZORB (immobilized lipase) cartridge — Hydrolyzing fats from enteral formula, ex vivo, with in-line enteral feed RELiZORB (immobilized lipase) cartridge
Other: Impact Peptide 1.5 — Impact Peptide 1.5 at a volume of administration from 500 mL to 1,000 mL per enteral feeding
  Other Names: Enteral Formula

SUMMARY:
Protocol 0000498: Multicenter, open label study to evaluate the effect of sustained RELiZORB (immobilized lipase) cartridge use during enteral feeding on fat absorption, as well as safety and tolerability of sustained RELiZORB use, in patients with cystic fibrosis and exocrine pancreatic insufficiency.

DETAILED DESCRIPTION:
Study Entry (Day -14): Baseline blood samples collected for plasma and erythrocyte concentrations of docosahexaenoic acid (DHA) and eicosapentaenoic (EPA). Baseline characteristics collected included BMI and cystic fibrosis related diabetes.

Observation Period (Day -14 to Day -8): Subjects followed their usual enteral nutrition regimen with pancreatic enzyme replacement therapy (PERT).

Run-in Period (Day -7 to Day -1): Subjects used Peptamen 1.5 enteral formula at their normal volume of administration from 500 mL to 1,000 mL per feeding with usual PERT regimen.

Treatment Period (Day 0 to Day 90): Subjects used Impact Peptide 1.5 up to a maximum volume of 1,000 mL per feeding with RELiZORB for the 90 day treatment period. Blood screening measurements were repeated at start of treatment period (Day 0), Day 30, Day 60 and Day 90. PERT use with enteral feedings was prohibited. Safety and tolerability were assessed with GI symptom diaries and systematic assessments of adverse events and unanticipated adverse device effects.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of cystic fibrosis
2. Documented history of exocrine pancreatic insufficiency
3. Enteral formula use a minimum of 4x/week, using PERT, consuming an unrestricted fat diet, and willing to use Peptamen 1.5 and Impact Peptide 1.5
4. Written informed consent or assent.

Exclusion Criteria:

1. Uncontrolled diabetes mellitus
2. Signs and symptoms of liver cirrhosis or portal hypertension
3. Lung or liver transplant
4. Active cancer currently receiving cancer treatment
5. Crohn's or celiac disease, infectious gastroenteritis, sprue, lactose intolerance, inflammatory bowel disease

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhumalli Sarkar, MD, PhD, Study Director — Alcresta Therapeutics, Inc.
Locations (10):
- United States (10):
  - Joe DiMaggio Children's Hospital / Memorial Healthcare System, Hollywood, Florida
  - St. Luke's CF Center of Idaho, Boise, Idaho
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Maine Medical Center, Portland, Maine
  - Helen DeVos Children's Hospital CF Care Center, Grand Rapids, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital / Saint Louis University, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted through Cystic Fibrosis Care Centers.
Pre-assignment Details: 7-day Observation Period: Maintain usual enteral feeding (EF) regimen. 7-day Run-in period: Maintain usual EF volume up to a max of 1000 mL using standard formula for at least 5 days.
  49 subjects signed consent; 5 screen failed; 44 started the observation period; 39 completed observation and run-in periods entering the treatment period.
Groups:
- Single Arm: Open Label: 49 subjects signed consent and were screened for the study. 44 subjects were eligible at time of screening. 39 subjects entered the treatment period.
Period: Overall Study
Arm/Group | Single Arm: Open Label
Started | 44
Enrolled | 44
Treated | 39
Completed | 36
Not Completed | 8
Not completed — Adverse Event | 4
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 1
Not completed — G-tube came out | 1
Not completed — Non-compliant use of PERT | 1

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: Open Label: RELiZORB cartridge and Impact Peptide 1.5 with enteral feeding 500 mL to 1,000 mL per enteral feeding for a period of 90 days.
  RELiZORB: Novel enteral feeding in-line digestive enzyme cartridge
  Impact Peptide 1.5: Impact Peptide 1.5 at a volume of administration from 500 mL to 1,000 mL per enteral feeding
Arm/Group | Single Arm: Open Label
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 37
  More than one race | 0
  Unknown or Not Reported | 0
Erythrocyte omega-3 index % [Mean (Standard Deviation); unit: % of omega-3 index of RBC membrane] — Population: ITT was 39, missing sample data due to one subject discontinuing prior Visit 3 therefore analysis population: N=38
  Erythrocyte omega-3 index % measures erythrocyte membrane composition (%) of DHA+EPA.
  % of omega-3 index of RBC membrane
    number analyzed (Participants) | 38
    (all) | 4.43 (2.05)
BMI [Mean (Standard Deviation); unit: weight (kg) / [height (m)]2] — BMI formula: weight (kg) / [height (m)]2
  weight (kg) / [height (m)]2 | 17.7 (1.8)
Cystic fibrosis related diabetes [Count of Participants; unit: Participants]
  Cystic fibrosis related diabetes | 9
  Non-cystic fibrosis related diabetes | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Erythrocyte Omega-3 Index % (DHA+EPA)
Description: Change from baseline Day 0 to Day 90 of erythrocyte tissue composition % of the omega-3 index
Time Frame: Day 0 to Day 90
Population: Intent to treat population = 39 subjects who received at least one exposure to RELiZORB. Analysis group is 38 due to one subject discontinuing prior to Visit 3.
Measure: Least Squares Mean (Standard Error); unit: percentage of omega-3 composition
Groups:
- RELiZORB Cartridge With Standard Enteral Formula: Patients with exocrine pancreatic insufficiency, age 5 and older, all sexes who have an enteral feeding a minimum of 4 times per week.
Arm/Group | RELiZORB Cartridge With Standard Enteral Formula
Number analyzed (Participants) | 38
percentage of omega-3 composition | 5.01 (0.40)

2. Secondary Outcome: Unanticipated Adverse Device Effects (UADE)
Description: A UADE is analogous to a serious adverse event (SAE), defined as an AE, occurring at any exposure to the therapeutic agent, that results in any of the following outcomes: death, life-threatening AE, inpatient hospitalization or prolonged existing hospitalization, a persistent or significant disability or incapacity or a congenital anomaly/birth defect.
Time Frame: RELiZORB Treatment Period (Day 0-Day 90): 90 days with additional 30 days of follow up.
Population: Total ITT population (n=39)
Measure: Number; unit: participants
Groups:
- RELiZORB Treatment Period (Day 0 - Day 90): All subjects who entered the RELiZORB Treatment period and received at least one treatment with the study device. 39 subjects entered treatment period of EF with RELiZORB.
Arm/Group | RELiZORB Treatment Period (Day 0 - Day 90)
Number analyzed (Participants) | 39
participants
  Patients with at least one UADE | 10
  Infections and Infestation | 2
  Respiratory, Thoracic, and Mediastinal | 8

3. Secondary Outcome: Changes in Plasma Concentration Total DHA+EPA
Description: Changes in plasma concentration total DHA+EPA from baseline (Day 0 to Day 90).
Time Frame: RELiZORB Treatment Period (Day 0-Day 90): 90 days
Population: All subjects who entered the RELiZORB Treatment period, received at least one treatment with the study device and completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of total plasma concentration
Groups:
- RELiZORB Treatment Period (Day 0 - Day 90): All subjects who entered the treatment period and received at least one exposure to RELiZORB.
Arm/Group | RELiZORB Treatment Period (Day 0 - Day 90)
Number analyzed (Participants) | 36
percentage of total plasma concentration | 93.73 [69.50 to 117.96]

4. Secondary Outcome: Erythrocyte Composition (%) of DHA
Description: Changes over time in erythrocyte composition (%) for total DHA in ITT population (n=39)
Time Frame: RELiZORB Treatment Period (Day 0-Day 90): 90 days
Population: ITTT
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of RBC composition
Arm/Group | RELiZORB Treatment Period (Day 0 - Day 90)
Number analyzed (Participants) | 39
percentage of RBC composition | 3.28 [2.74 to 3.82]

5. Secondary Outcome: Erythrocyte Composition (%) of EPA
Description: Changes over time in erythrocyte composition (%) for EPA in ITT population
Time Frame: RELiZORB Treatment Period (Day 0-Day 90): 90 days
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of RBC composition
Arm/Group | RELiZORB Treatment Period (Day 0 - Day 90)
Number analyzed (Participants) | 39
percentage of RBC composition | 1.73 [1.32 to 2.14]

6. Secondary Outcome: Erythrocyte Composition (%) Ratio of n6/n3 Fatty Acids
Description: Change from baseline to Day 90 in n6/n3 ratio in erythrocytes
Time Frame: RELiZORB Treatment Period (Day 0-Day 90): 90 days
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of RBC composition
Arm/Group | RELiZORB Treatment Period (Day 0 - Day 90)
Number analyzed (Participants) | 39
percentage of RBC composition | -2.51 [-2.94 to -2.09]

7. Secondary Outcome: Plasma Composition (%) Ratio of n6/n3 Fatty Acids.
Description: Change over time in n6/n3 ratio in plasma in the ITT population
Time Frame: RELiZORB Treatment Period (Day 0-Day 90): 90 days
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of total plasma concentration
Arm/Group | RELiZORB Treatment Period (Day 0 - Day 90)
Number analyzed (Participants) | 39
percentage of total plasma concentration | -6.29 [-7.85 to -4.73]

8. Other Pre Specified Outcome: GI Symptoms
Description: GI symptoms recorded in GI diaries by subject and/or caregiver.
Time Frame: Observation, Baseline and RELiZORB Treatment periods (Day -14 to Day 90): 104 days with additional 30 days of follow up.
Population: All subjects who entered the RELiZORB Treatment Period and received at least one treatment with RELiZORB.
Measure: Count of Participants; unit: Participants
Groups:
- Safety Population: All subjects who entered the RELiZORB Treatment period and received at least one treatment with the study device. 39 subjects entered treatment period of EF with RELiZORB.
Arm/Group | Safety Population
Number analyzed (Participants) | 39
Participants
  Study Entry | 23
  End of Study | 12

ADVERSE EVENTS:
Time Frame: Adverse event data collected and reported for 14 days during the Observation and Run-in periods. Adverse event data collected and reported for 120 days for the RELiZORB period.
Description: Adverse event data were collected from study entry at day -14 to end of study (Day -14 through 90). Follow up of events present at end of study/termination continued for an additional 30 days after completion of study.
Groups:
- Observation and Run-in Period (Day -14 to Day -1): This 14 day period was comprised of 7 day Observation period followed by 7 day Run-in period. 44 subjects were enrolled of which 39 proceeded to treatment period of EF with RELiZORB.
- RELiZORB Treatment Period (Day 0 - Day 90): Safety population is defined as all subjects who entered the RELiZORB Treatment period and received at least one treatment with the study device. 39 subjects entered treatment period of EF with RELiZORB.
Arm/Group | Observation and Run-in Period (Day -14 to Day -1) | RELiZORB Treatment Period (Day 0 - Day 90)
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/39
Serious Adverse Events (participants affected / at risk) | 2/44 | 0/39
Other Adverse Events (participants affected / at risk) | 4/44 | 23/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observation and Run-in Period (Day -14 to Day -1) (N=44) | RELiZORB Treatment Period (Day 0 - Day 90) (N=39)
Infectious colitis (Infections and infestations) | 1 (1) | 0 (0)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observation and Run-in Period (Day -14 to Day -1) (N=44) | RELiZORB Treatment Period (Day 0 - Day 90) (N=39)
Vomiting (Gastrointestinal disorders) | 4 (6) | 0 (0)
Pulmonary function decreased (Investigations) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (9)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 10 (12)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Ear infection (Infections and infestations) | 0 (0) | 2 (2)
Forced expiratory volume decreased (Investigations) | 0 (0) | 2 (2)
Vitamin D decrease (Investigations) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Patient GI symptom diary: recall method using unvalidated tool. Patients were allowed to eat normal diet during the day, hence the amount of LCPUFA that was measured in the plasma is not the sole reflection of the device use only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication by the PI of any data from this study is strictly prohibited without consent from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-03-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT02750501/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT02750501/SAP_001.pdf